CLINICAL TRIAL: NCT00982436
Title: A Pilot Study to Evaluate Response to Neoadjuvant Chemotherapy With Cisplatin and Docetaxel Followed by Chemoradiation Therapy With Carboplatin in Stage IV Non-metastatic Head and Neck Cancer
Brief Title: Neoadjuvant Cisplatin/Docetaxel (CDDP/TXT) and Chemoradiation for Head and Neck Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Steven Grunberg, Professor of Medicine, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VCC 0905
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Head and Neck Neoplasms
Keywords: Combined Modality Therapy; Neoadjuvant Therapy; Head and neck neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Radiotherapy; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Neoadjuvant/Concomitant Chemoradiation (Experimental): Three cycles of docetaxel/carboplatin neoadjuvant chemotherapy followed by chemoradiotherapy for 7 weeks with weekly carboplatin
  Interventions: Drug: Docetaxel/cisplatin; Radiation: Radiotherapy; Drug: Carboplatin

INTERVENTIONS:
Drug: Docetaxel/cisplatin — Docetaxel 75 mg/m2 intravenous every 3 weeks for 3 cycles Cisplatin 75 mg/m2 intravenous every 3 weeks for 3 cycles
  Other Names: Taxotere; Platinol
Radiation: Radiotherapy — 70 Gy in 35 fractions to gross tumor and lymph node metastases
  Other Names: Radiation therapy
Drug: Carboplatin — Carboplatin AUC 1.5 intravenous weekly during radiotherapy
  Other Names: Paraplatin

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of neoadjuvant chemotherapy (chemotherapy given before radiotherapy) using cisplatin and docetaxel, followed by carboplatin given at the same time as radiotherapy in the treatment of locally advanced head and neck cancer.

DETAILED DESCRIPTION:
Chemoradiotherapy has become the standard of care for patients with unresectable head and neck cancer, but there can be substantial added toxicity with chemoradiotherapy compared to radiation therapy alone. Neoadjuvant therapy with cisplatin / 5-fluorouracil has demonstrated activity in this disease, and taxanes appear to improve response further. Docetaxel / cisplatin / 5-fluorouracil has been shown to be a highly active regimen. However, with the potential added toxicities of neoadjuvant chemotherapy, it is important to minimize toxicity while maintaining efficacy. Chemotherapeutic agents that are DNA cycle-specific like 5-fluorouracil are more stomatotoxic than those that are cell phase non-specific. Of note, several studies have suggested that docetaxel and cisplatin is a highly active combination when used for advanced disease or as neoadjuvant therapy .

This study will therefore test the efficacy of neoadjuvant chemotherapy with cisplatin and docetaxel without 5-fluorouracil followed by chemoradiotherapy with carboplatin to determine whether promising response rates with modest toxicity can be achieved. Carboplatin will be used as the radiosensitizing agent during chemoradiotherapy to reduce nephrotoxicity and neurotoxicity as compared to further treatment with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven locoregional Stage 4 squamous cell carcinoma of the oral cavity, larynx, oropharynx or hypopharynx
* Measurable or evaluable disease
* No distant metastases
* Tumor should be surgically unresectable for cure or resection is considered inadvisable
* Age > 18 years
* ECOG performance status 0, 1 or 2
* Life expectancy > 2 months
* Patients must have adequate organ and marrow function as defined below:

  * Leukocytes > 3,000/mm3
  * Absolute neutrophil count > 1,500/mm3
  * Platelets > 100,000/mm3
  * Hemoglobin > 10.0g/dL
  * Total Bilirubin <= institutional upper limit of normal
  * Aspartate aminotransferase < 2.5 X institutional upper limit of normal
  * Alanine aminotransferase < 2.5 X institutional upper limit of normal
  * Alkaline phosphatase < 2.5 X institutional upper limit of normal
  * Creatinine <= institutional upper limit of normal OR creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine > institutional upper limit of normal
* Signed informed consent
* Women of child-bearing potential and men must be willing and able practice adequate contraception prior to study entry and for the duration of study treatment

Exclusion Criteria:

* Previous chemotherapy for this malignancy
* Previous radiotherapy to head and neck region
* Other malignancy within last 5 years except for non-melanoma skin cancer
* Uncontrolled intercurrent illness that would prevent delivery of protocol therapy
* Peripheral neuropathy > Grade 2
* Hypercalcemia
* Patient is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Response rate to neoadjuvant chemotherapy with docetaxel/cisplatin, followed by chemoradiotherapy in locally advanced squamous head and neck cancer | 6 months after initiation of therapy

SECONDARY OUTCOMES:
Response rate to neoadjuvant chemotherapy with docetaxel/cisplatin in locally advanced squamous head and neck cancer | 3 months after initiation of therapy
Response rate to chemoradiotherapy in locally advanced squamous head and neck cancer | 6 months after initiation of therapy
Toxicity of neoadjuvant chemotherapy with docetaxel/cisplatin, followed by chemoradiotherapy in locally advanced squamous head and neck cancer | Every 3 weeks for 6 months (during therapy)
Progression free survival after neoadjuvant chemotherapy with docetaxel/cisplatin, followed by chemoradiotherapy in locally advanced squamous head and neck cancer | Every 6 months
Overall survival after neoadjuvant chemotherapy with docetaxel/cisplatin, followed by chemoradiotherapy in locally advanced squamous head and neck cancer | Every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Grunberg, MD, Principal Investigator — University of Vermont/Feltcher Allen Health Care
Locations (3):
- United States (3):
  - Mountainview Medical Center, Berlin Corners, Vermont
  - Fletcher Allen Health Care, Burlington, Vermont
  - Vermont Center for Cancer Medicine, Colchester, Vermont